CLINICAL TRIAL: NCT04223245
Title: A Comparison Of Home Exercises With Multimodal Real-time Sensory Feedback To The Same Exercise Program With No Enhanced Feedback on Walking Automaticity in People With Parkinson Disease.
Brief Title: A Home Program Using Multimodal Sensory Feedback for People With Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regis University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1008713-3
Record Dates: First submitted 2019-12-02; First posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Parkinson Disease
Keywords: multimodal; real-time feedback; automaticity; gait; balance
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Single blind randomized trial with 2 groups
Who Masked: Outcomes Assessor
Masking Description: blinded to subject group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise+MMSF (Experimental): Group of PWPD who performed a base exercise program of speed and large amplitude stepping and standing balance exercises with Multimodal real-time sensory feedback
  Interventions: Behavioral: exercise+multi-modal sensory feedback (MMSF)
- exercise only (Active Comparator): Group PWPD who did the same exercise program without MMSF
  Interventions: Behavioral: Exercise only

INTERVENTIONS:
Behavioral: exercise+multi-modal sensory feedback (MMSF) — home program of 3 stepping exercises and 3 balance exercises with progression of speed, step distance and reduced vision. Real-time sensory feedback during ex. using ankle, wrist wts., laser on chest and mat with footpads and clickers (auditory feedback during stepping)
  Arms: exercise+MMSF
Behavioral: Exercise only — 3 stepping and 3 balance exercises which are to progress in speed and distance of movement as well as progress to eyes closed while performing.
  Arms: exercise only

SUMMARY:
People with Parkinson Disease (PWPD) have significant problems with velocity, safety and dual tasking during walking that may be secondary to poor automaticity. Sensory functions, especially visual dependence and proprioceptive integration are critical for efficient walking and are often impaired. This home program compares the use of multimodal sensory feedback during stepping and balance exercises in PWPD to a group without the sensory feedback performing the same basic exercises.

DETAILED DESCRIPTION:
Parkinson disease impairs motor and sensory functions. Automaticity of gait is lost increasing the use of higher center control of walking, leading to cognitive fatigue, slower movement and motor errors. People with Parkinson disease (PWPD) improve motor performance when external sensory cues, which bypass the faulty basal ganglia, are used during interventions. Enhancing proprioceptive, visual and vestibular cues that are critical for walking has the potential to improve gait and decrease cognitive fatigue by restoring automaticity.

This is a single-blinded randomized controlled study with repeated measures to evaluate the effects of a home exercise program with or without the addition of multi-modal sensory feedback (MMSF) in real-time on automaticity of gait and balance. PWPDs are randomly assigned to one of 2 home exercise groups. There are two 6 week exercise sessions with a 6 week of no exercises inter-spaced between them. The exercises promote rapid and large movement in stepping activities, balance using self-perturbation through single, leg swings and standing on a compliant surface for sensory re-weighting. People in the experimental group perform the program with real-time with MMSF. Participants are to progress exercises in speed and distance as well as performing with eyes closed to improve proprioceptive processing and automaticity.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of Parkinson Disease
* A score of 26 or higher on the Mini-Mental Status Exam
* Able to stand from sitting and take 5 steps without assistance
* People who have been on the same dosages of medication for PD for 3 weeks or longer

Exclusion Criteria:

* Participating in an exercise program for less than 3 months
* Plans to change a current exercise program during the study
* Changes in medications that affect PD or its sequelea

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2019-03-08 (Actual)

PRIMARY OUTCOMES:
Changes in temporalspatial components of Gait | baseline before exercise training, 6 weeks, 12 weeks and 18 weeks after initiation of exercise
  temporal and spacial components of gait measured with Gaitrite Mat
changes in balance | baseline before exercise training, 6 weeks, 12 weeks and 18 weeks after initiation of exercise
  single leg stance time, time standing on foam eyes closed, Mini-BESTest
Change in cognitive attention needed for gait | Baseline, 6 weeks, 12 weeks and 18 weeks after initiation of exercise
  3 meter walk test performed at comfortable gait speed once and repeated while subtracting 3s from 100 to assess cognitive attention needed for walking tasks (automaticity)
Change in perceived difficulty during gait and ADLs, | Baseline, 6 weeks, 12 weeks and 18 weeks after initiation of exercise
  Parkinson Disease Questionnaire (PDQ-39)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A Winkler, PT, DSc, Principal Investigator — Regis University, 3333 Regis Blvd , Denver, Co 80221
Locations (1):
- Regis University, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No